CLINICAL TRIAL: NCT03135548
Title: Multi-center, Double-blind, Randomised, Placebo-controlled, Phase IIa Study to Investigate Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacogenomics of Multiple Intravenous Doses of BI 655130 in Patients With Palmoplantar Pustulosis (PPP)
Brief Title: Initial Dosing of BI 655130 in Palmoplantar Pustulosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0015; 2016-004573-40 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spesolimab (low dose) (Experimental)
  Interventions: Drug: Spesolimab (low dose)
- Spesolimab (high dose) (Experimental)
  Interventions: Drug: Spesolimab (high dose)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spesolimab (low dose) — 12 weeks treatment
  Arms: Spesolimab (low dose)
Drug: Placebo — 12 weeks treatment
  Arms: Placebo
Drug: Spesolimab (high dose) — 12 weeks treatment
  Arms: Spesolimab (high dose)

SUMMARY:
The primary objective of this trial is to investigate the safety and efficacy of BI 655130 in patients with PPP following multiple intravenous administrations compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 to 65 years of age at screening.
* Palmoplantar Pustulosis
* Further inclusion criteria apply

Exclusion Criteria:

* Presence or known history of anti- Tumor necrosis factor (TNF)-induced Palmoplantar Pustulosis (PPP)-like disease.
* Active or latent tuberculosis
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Canada (3):
  - Dr. Irina Turchin PC Inc., Fredericton, New Brunswick
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
- Denmark (3):
  - Aarhus University Hospital, Skejby, Aarhus
  - Gentofte Hospital, Hellerup
  - Bispebjerg og Frederiksberg Hospital, København NV
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - TFS Trial Form Support GmbH, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
- Italy (2):
  - Ospedale San Giovanni di Dio, Cagliari
  - Pol. Universitario Tor Vergata, Roma
- Spain (3):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Ramón y Cajal, Madrid
- Sweden (2):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Karolinska Univ. sjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, placebo-controlled, parallel-design trial to investigate the safety and efficacy of BI 655130 in patients with Palmoplantar Pustulosis (PPP) following multiple intravenous administrations of either low dose or high dose compared with placebo.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensured that all participants met all inclusion/exclusion criteria. Participants were not to be randomised to trial treatment if any one of the specific entry criteria were not met.
Groups:
- BI 655130 Low Dose: Participants were administered low dose of BI 655130 solution for infusion intravenously every 4 weeks at Day 1, 29, 57 and 85 until 12 weeks.
- BI 655130 High Dose: Participants were administered high dose of BI 655130 solution for infusion intravenously every 4 weeks at Day 1, 29, 57 and 85 until 12 weeks.
- Placebo Matching to BI 655130: Participants were administered placebo matching to BI 655130 solution for infusion intravenously every 4 weeks at Day 1, 29, 57 and 85 until 12 weeks.
Period: Overall Study
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130
Started (Started are randomised/treated) | 19 | 19 | 21
Completed | 14 | 15 | 18
Not Completed | 5 | 4 | 3
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Other than listed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): SAF included all randomised patients who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130 | Total
Number analyzed (Participants) | 19 | 19 | 21 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (7.7) | 49.4 (11.3) | 46.3 (11.7) | 50.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 17 | 49
  Male | 3 | 3 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 17 | 16 | 20 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 18 | 19 | 19 | 56
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Palmoplantar (pp) Pustular Psoriasis Area and Severity Index 50 (PASI) (ppPASI50) at Week 16
Description: Percentage of participants who achieved 50% reduction in ppPASI score was assessed by ppPASI50.
  ppPASI is modification of PASI score and an investigator assessment of the extent and severity of pustular and plaque lesions on the palms and soles presenting in PPP participants. This tool provides a numeric scoring for participants overall PPP disease state, ranging from 0 to maximum 72, where 0 corresponds to no signs of psoriasis. It is a linear combination of the percent of surface area of skin that is affected on the palms and soles and the severity of Erythema (E), Pustules (P) (total), and scaling (Desquamation (D)). Missing values for severity or area of involvement were not imputed.
  ppPASI was calculated as a weighted sum of the scores obtained for E, P, D and Area affected (in%) (where area assessed is glabrous skin on the palms/ soles) (A): [(E+P+D) x A x 0.2 (right palm)] + [(E+P+D) x A x 0.2 (left palm)] + [(E+P+D) x A x 0.3 (right sole)] + [(E+P+D) x A x 0.3 (left sole)].
Time Frame: Week 16
Population: Full analysis set (FAS): FAS included all patients in the Safety analysis set (SAF) (SAF included all randomised patients who received at least one dose of study drug) who had a baseline measurement available for the primary endpoint. Patients from FAS with no response imputation (NRI) were included for analysis of this endpoint. (FAS (NRI))
Measure: Number; unit: Percentage of participants (%)
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130
Number analyzed (Participants) | 19 | 19 | 21
Percentage of participants (%) | 31.6 | 31.6 | 23.8
Statistical Analysis 1: Comparison: BI 655130 Low Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Wilson/Newcombe; 95% confidence intervals (CI) are calculated using the method of Wilson/Newcombe; Risk Difference (RD) = 0.078, 95% CI 2-sided [-0.190 to 0.338] — Unadjusted absolute risk difference versus placebo was calculated as the difference in the observed proportion of patients with ppPASI50 at Week 16 for each treatment scenario, for the FAS
Statistical Analysis 2: Comparison: BI 655130 High Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Wilson/Newcombe; 95% CIs are calculated using the method of Wilson/Newcombe; Risk Difference (RD) = 0.078, 95% CI 2-sided [-0.190 to 0.338] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants With Drug-related Adverse Events (AEs)
Description: Number of participants with drug-related AEs are presented.
Time Frame: From first drug administration until 16 weeks after the last drug administration, up to 32 weeks.
Population: Safety analysis set (SAF): This set included all randomised patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130
Number analyzed (Participants) | 19 | 19 | 21
Participants | 8 | 8 | 9

3. Secondary Outcome: Percentage of Participants With Palmoplantar Pustular Psoriasis Area and Severity Index 75 (ppPASI75) at Week 16
Description: Percentage of participants who achieved >75% reduction in ppPASI score was assessed by ppPASI75.
  ppPASI is modification of PASI score and an investigator assessment of the extent and severity of pustular and plaque lesions on the palms and soles presenting in PPP participants. This tool provides a numeric scoring for participants overall PPP disease state, ranging from 0 to maximum 72, where 0 corresponds to no signs of psoriasis. It is a linear combination of the percent of surface area of skin that is affected on the palms and soles and the severity of Erythema (E), Pustules (P) (total), and scaling (Desquamation (D)). Missing values for severity or area of involvement were not imputed.
  ppPASI was calculated as a weighted sum of the scores obtained for E, P, D and Area affected (in%) (where area assessed is glabrous skin on the palms/ soles) (A): [(E+P+D) x A x 0.2 (right palm)] + [(E+P+D) x A x 0.2 (left palm)] + [(E+P+D) x A x 0.3 (right sole)] + [(E+P+D) x A x 0.3 (left sole)].
Time Frame: Week 16
Population: FAS (NRI)
Measure: Number; unit: Percentage of participnats (%)
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130
Number analyzed (Participants) | 19 | 19 | 21
Percentage of participnats (%) | 0.0 | 21.1 | 9.5
Statistical Analysis 1: Comparison: BI 655130 Low Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Wilson/Newcombe; 95% CIs are calculated using the method of Wilson/Newcombe; Risk Difference (RD) = -0.095, 95% CI 2-sided [-0.289 to 0.086] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 655130 High Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Wilson/Newcombe; 95% CIs are calculated using the method of Wilson/Newcombe; Risk Difference (RD) = 0.115, 95% CI 2-sided [-0.116 to 0.348] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percent Change From Baseline in the ppPASI at Week 16
Description: The percentage change in the ppPASI score from Baseline to Week 16 was measured.
  ppPASI is modification of PASI score and an investigator assessment of the extent and severity of pustular and plaque lesions on the palms and soles presenting in PPP participants. This tool provides a numeric scoring for participants overall PPP disease state, ranging from 0 to maximum 72, where 0 corresponds to no signs of psoriasis. It is a linear combination of the percent of surface area of skin that is affected on the palms and soles and the severity of Erythema (E), Pustules (P) (total), and scaling (Desquamation (D)). Missing values for severity or area of involvement were not imputed.
  ppPASI was calculated as a weighted sum of the scores obtained for E, P, D and Area affected (in%) (where area assessed is glabrous skin on the palms/ soles) (A): [(E+P+D) x A x 0.2 (right palm)] + [(E+P+D) x A x 0.2 (left palm)] + [(E+P+D) x A x 0.3 (right sole)] + [(E+P+D) x A x 0.3 (left sole)].
Time Frame: Baseline and Week 16
Population: Patients from FAS with observed cases (OC) were included for analysis of this endpoint. (FAS (OC))
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130
Number analyzed (Participants) | 15 | 14 | 15
Unit on scale | -32.74 (38.52) | -45.80 (27.00) | -39.97 (32.94)
Statistical Analysis 1: Comparison: BI 655130 Low Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Student's t-distribution; CIs were based on Student's t-distribution; Mean Difference (Final Values) = 7.24, 95% CI 2-sided [-20.01 to 34.48]
Statistical Analysis 2: Comparison: BI 655130 High Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Student's t-distribution; CIs were based on Student's t-distribution; Mean Difference (Final Values) = -5.82, 95% CI 2-sided [-28.35 to 16.70]

5. Secondary Outcome: Percentage of Participants Achieving Treatment Success (Treatment Success Defined as Achieving a Clinical Response of 0 or 1=Clear/Almost Clear) Via Palmoplantar Pustulosis Physicians Global Assessment (pppPGA) at Week 16
Description: pppPGA was relied on the participant's overall skin lesions status on the lesions of the most severely affected palmoplantar surface of the palms and sole was assessed by investigator as clear (0), almost clear (1), mild (2), moderate (3) and severe (4) at week 16.
  Score Wording were:
  0 = Clear = No signs of PPP; no scaling or crusts or pustule remains.
  1. = Almost clear = Slight scaling and/or erythema and / or slight crusts; very few new (yellow) and / or old (brown) pustules.
  2. = Mild = Scaling and/or erythema and/or crusts; visible new (yellow) and/or old (brown) pustules of limited number and extent.
  3. =Moderate = Prominent scaling and/or erythema and / or crusting; prominent new (yellow) and / or old (brown) pustules covering most of the area involved.
  4. =Severe = Severe scaling and/or erythema and / or crusting; numerous new (yellow) or old (brown) pustules with and/or without major conflence covering the entire area of at least 2 palmoplantar surfaces.
Time Frame: Week 16
Population: FAS (NRI)
Measure: Number; unit: Percentage of participants (%)
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130
Number analyzed (Participants) | 19 | 19 | 21
Percentage of participants (%) | 0.0 | 15.8 | 14.3
Statistical Analysis 1: Comparison: BI 655130 Low Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Wilson/Newcombe; 95% CIs are calculated using the method of Wilson/Newcombe; Risk Difference (RD) = -0.143, 95% CI 2-sided [-0.346 to 0.049]
Statistical Analysis 2: Comparison: BI 655130 High Dose vs Placebo Matching to BI 655130; Test type: Other — No formal hypothesis testing was performed in this trial; Wilson/Newcombe; 95% CIs are calculated using the method of Wilson/Newcombe; Risk Difference (RD) = 0.015, 95% CI 2-sided [-0.213 to 0.252]

ADVERSE EVENTS:
Time Frame: From first drug administration until 16 weeks after the last drug administration, up to 32 weeks.
Description: Analysis set for safety presentation was Safety analysis set (SAF). SAF included all randomised patients who received at least one dose of study drug.
Arm/Group | BI 655130 Low Dose | BI 655130 High Dose | Placebo Matching to BI 655130
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19 | 1/21
Other Adverse Events (participants affected / at risk) | 17/19 | 17/19 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655130 Low Dose (N=19) | BI 655130 High Dose (N=19) | Placebo Matching to BI 655130 (N=21)
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655130 Low Dose (N=19) | BI 655130 High Dose (N=19) | Placebo Matching to BI 655130 (N=21)
Nasopharyngitis (Infections and infestations) | 5 | 8 | 8
Urinary tract infection (Infections and infestations) | 1 | 3 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Alcohol intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 4 | 6 | 7
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Bundle branch block (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Administration site extravasation (General disorders) | 1 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03135548/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03135548/SAP_001.pdf